CLINICAL TRIAL: NCT01381471
Title: Fluticasone Propionate-salmeterol Combination Adherence in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 113865
Record Dates: First submitted 2011-06-23; First posted 2011-06-27 (Estimated); Results first posted 2012-03-07 (Estimated); Last update posted 2012-03-29 (Estimated); Status verified 2012-02

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- COPD: Patients with a diagnosis code of COPD
  Interventions: Drug: fluticasone propionate/salmeterol xinafoate combination

INTERVENTIONS:
Drug: fluticasone propionate/salmeterol xinafoate combination — fluticasone propionate/salmeterol xinafoate combination
  Other Names: Advair (TM)

SUMMARY:
The specific aim of this study is to describe 1 year Advair dispensing rates for patients with COPD, and to measure the association between Advair adherence and healthcare utilization (e.g. emergency room visits and inpatient admissions, etc.). To compare the risk of a COPD exacerbation (moderate or severe) during a 3-month follow-up period between patients thqat are adherent versus those that are not.

ELIGIBILITY:
INCLUSION CRITERIA

* at least one pharmacy claim for Advair (any strength; Diskus or MDI) during the index year (July 1, 2005 through June 30, 2006).
* Continuous medical and pharmacy eligibility for the 12 month Pre-Index year and the 12 month Index year (referred to as the 24 month Observation Period), and the 3 month Post-Index period (referred to as the Outcome Period).
* At least one medical claim with a diagnosis (either primary or secondary) of COPD (ICD-9 code 490.xx, 491.xx, 492.xx, and 496), AND at least 1 pharmacy claim for an Anticholinergic medication, both occurring during the12 month pre-index period.
* At least 40 years old at index date.

EXCLUSION CRITERIA

* any medical claim (ever) with a primary or secondary diagnosis of cystic fibrosis (ICD-9 code 277.0x).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 40 years of age or older with at least one pharmacy claim for FSC during the index date range (July 1, 2005 through June 30, 2006). An index date was designated as the date of the first pharmacy claim for FSC. Patients were also required to have continuous medical and pharmacy eligibility for the 12 month pre-Index year and the 12 month Index year (referred to as the 24 month observation period), and the 3 month post-Index outcome period (referred to as the outcome period). Eligible patients were further required to have at least one medical claim with a diagnosis (either primary or secondary) of COPD (ICD-9-CM code 490.xx, 491.xx, 492.xx, and 496), AND at least 1 pharmacy claim for an anticholinergic medication, both occurring during the12 month pre-index period.
Sampling Method: Non-Probability Sample
Enrollment: 11060 (Actual)
Dates: Start 2009-08; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were not recruited or enrolled in this study. This study is a retrospective observational study. Data from medical records or insurance claims databases are anonymized and were used to develop a cohort. All diagnoses and treatments are recorded in the course of routine medical practice.
Groups:
- Fluticasone Propionate/Salmeterol (FSC): Participants age 40 or older with at least one pharmacy claim for FSC, at least one medical claim with a primary or secondary diagnosis of Chronic Obstructive Pulmonary Disease (COPD) (International Classification of Disease, 9th Revision [ICD-9], Clinical Modification codes 490.xx, 491.xx, 492.xx, or 496.xx), and at least one pharmacy claim for an anticholinergic medication but no diagnosis for cystic fibrosis (ICD-9 = 277.0x)
Period: Overall Study
Arm/Group | Fluticasone Propionate/Salmeterol (FSC)
Started | 11060
Completed | 11060
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Fluticasone Propionate/Salmeterol (FSC): Participants age 40 or older with at least one pharmacy claim for FSC, at least one medical claim with a primary or secondary diagnosis of Chronic Obstructive Pulmonary Disease (COPD) (International Classification of Disease, 9th Revision [ICD-9], Clinical Modification [ICD-9] codes 490.xx, 491.xx, 492.xx, or 496.xx), and at least one1 pharmacy claim for an anticholinergic medication but no diagnosis for cystic fibrosis (ICD-9 = 277.0x)
Arm/Group | Fluticasone Propionate/Salmeterol (FSC)
Number analyzed (Participants) | 11060
Age Continuous [Mean (Standard Deviation); unit: Years] | 61.6 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6103
  Male | 4957
Number of Participants with the Indicated Level of Adherence to FSC [Number; unit: participants] — Adherence levels were defined by the number of pharmacy claims for each participant in the year following the index date (an FSC claim from (July 1, 2005 to June 30, 2006). Three or fewer claims for FSC was considered low adherence, medium adherence was defined as 4 to 8 claims, and high adherence was defined as nine or more pharmacy claims.
  participants
    Low adherence | 2726
    Medium adherence | 3479
    High adherence | 4855

OUTCOME MEASURES:

1. Primary Outcome: Mean Number of Pharmacy Claims by Participants During the Post-Index Period
Description: The mean number of pharmacy claims incurred by participants during the one-year post-index period was measured.
Time Frame: One Year
Population: Participants age 40 or older with at least one pharmacy claim for FSC, at least one medical claim with a primary or secondary diagnosis of COPD (ICD-9 codes 490.xx, 491.xx, 492.xx, or 496.xx), and at least one pharmacy claim for an anticholinergic medication but no diagnosis for cystic fibrosis (ICD-9 = 277.0x)
Measure: Mean (Standard Deviation); unit: pharmacy claims
Arm/Group | Fluticasone Propionate/Salmeterol (FSC)
Number analyzed (Participants) | 11060
pharmacy claims
  Albuterol Pharmacy Claims | 2.960 (4.627)
  Inhaled Corticosteriod Pharmacy Claims | 0.219 (1.092)
  Anticholinergic Pharmacy Claims | 5.491 (5.397)
  Theophylline Pharmacy Claims | 0.573 (2.188)
  Oral Corticosteriod Pharmacy Claims | 1.545 (2.727)
  Antibiotic Pharmacy Claims | 2.181 (2.743)

2. Primary Outcome: Mean Number of Healthcare Encounters Incurred by Participants During the Post-Index Period
Description: The mean number of outpatient office visits, inpatient visits, and emergency department visits incurred by participants during the one-year post-index period was measured.
Time Frame: One Year
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: healthcare encounters
Arm/Group | Fluticasone Propionate/Salmeterol (FSC)
Number analyzed (Participants) | 11060
healthcare encounters
  Outpatient Office Visits | 2.048 (2.918)
  Emergency Department Visits | 0.145 (0.788)
  Inpatient Visits | 0.078 (0.353)

ADVERSE EVENTS:
Description: This is a retrospective study of pre-existing medical record and/or health insurance claims data; all data are de-identified, and thus no assessments of Serious or Non-serious Adverse Events are possible.
Arm/Group | Fluticasone Propionate/Salmeterol (FSC)
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.